CLINICAL TRIAL: NCT05222529
Title: A Phase II, Double-blind, Randomized, Multiple Dose, Cross Over, Three-treatment, Three-period, Six Sequence Placebo Controlled Trial to Evaluate Efficacy, Pharmacokinetics (PK), Pharmacodynamics (PD) and Safety and Tolerability of Glycopyrronium (Bromide) in Children From 6 to Less Than 12 Years of Age With Asthma.
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Glycopyrronium (Bromide) in Children (6 to Less Than 12 Years) With Asthma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVM149C2201; 2021-004972-32 (EudraCT Number)
Record Dates: First submitted 2022-01-10; First posted 2022-02-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: Glycopyrronium, pediatric, asthma, Breezhaler, PK
MeSH Terms: conditions — Asthma | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigator staff, persons performing the assessments, data analysts and the Sponsor Clinical Trial Team (CTT) will remain blind to the identity of the treatment from the time of randomization until database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glycopyrronium 25μg (Experimental): Glycopyrronium 25μg for two weeks
  Interventions: Drug: Glycopyrronium bromide 25ug; Drug: Placebo; Drug: Glycopyrronium bromide 12.5ug
- Glycopyrronium 12.5μg (Experimental): Glycopyrronium 12.5μg for two weeks
  Interventions: Drug: Glycopyrronium bromide 25ug; Drug: Placebo; Drug: Glycopyrronium bromide 12.5ug
- Placebo (Placebo Comparator): Placebo for two weeks
  Interventions: Drug: Glycopyrronium bromide 25ug; Drug: Placebo; Drug: Glycopyrronium bromide 12.5ug

INTERVENTIONS:
Drug: Glycopyrronium bromide 25ug — 25μg Glycopyrronium bromide capsules for oral inhalation via Breezhaler
  Other Names: NVA237
Drug: Placebo — Placebo to Glycopyrronium bromide capsules for oral inhalation via Breezhaler
Drug: Glycopyrronium bromide 12.5ug — 12.5ug Glycopyrronium bromide capsules for oral inhalation via Breezhaler
  Other Names: NVA237

SUMMARY:
The purpose of this study is to characterize the bronchodilator effect, systemic exposure and safety/tolerability of two different doses of inhaled glycopyrronium, when compared to placebo. Outcome of this study will be used to determine the dose of inhaled glycopyrronium for the development of fixed dose combination indacaterol/mometasone/glycopyrronium (QVM149) for children aged 6 to less than 12 years old with moderate to severe asthma.

DETAILED DESCRIPTION:
The study design is a double-blind, placebo controlled, randomized sequence, three-treatment, three-period, six-sequence, cross-over multiple-dose study to evaluate efficacy, pharmacokinetics, pharmacodynamics, and safety and tolerability of glycopyrronium bromide (bromide) in children from 6 to less than 12 years of age with asthma with forced expiratory volume in one second (FEV1) ≥60% and ≤ 90% of the predicted normal value for the participant.

This study will consist of 4 phases: Screening, Run-in, Treatment and Follow-up.

After the screening phase, participants will enter the Run-in Phase to further assess eligibility and those participants that meet all eligibility criteria will be randomized. Study treatment will be administered in addition to background asthma LABA+ICS controller therapy (salmeterol xinafoate 50µg/fluticasone propionate 100µg) from entering the run-in period, through to the end of the treatment phase, including the 2 wash-out periods. Participants will be randomized to one of 6 different sequences with an equal (1:1:1:1:1:1) randomization ratio. The Treatment Phase will last 10 weeks, and every sequence is divided in three treatment periods: Glycopyrronium bromide 12.5 µg, Glycopyrronium bromide 25µg or matching placebo dry powder in capsules for inhalation, via Breezhaler. Each treatment period lasts 2 weeks and 2 consecutive treatment periods are separated by a 2-week wash-out period. Participants who discontinue their study treatment prematurely will be required to return to the clinic for an Early Termination Visit. 30 days after last treatment date, a final telephone contact must be conducted for safety follow-up.

The total duration of the trial for a participant (from screening to follow up) is approximately 20 weeks including safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of asthma for at least 6 months
* Signed informed consent by parent(s)/legal guardian(s) and assent by the pediatric participant (depending on local requirements)
* Participant on stable dose of inhaled low-to-medium dose ICS with one additional controller for at least 4 weeks prior to run-in
* Pre-Bronchodilator FEV1 ≥60% to ≤90% of predicted normal at beginning of Run-in and randomization. If FEV1 eligibility criteria are not met at -45min pre-dose of the End of Run-in (Visit 30), the visit can be rescheduled once within 5 days from the previous attempt.
* FEV1 reversibility, done using up to 4 puffs of SABA (up to 400μg salbutamol or 360μg albuterol) at Run-in visit (Visit 20): increase > and/or = 12% (performed according to American Thoracic Society (ATS)/European Respiratory Society (ERS) 2019 guidelines). All participants must perform a reversibility test at start of Run-in. If reversibility is not demonstrated at Run-in, it may be attempted at up to two ad hoc, unscheduled separate visits within 5 days from previous attempt. If reversibility is still not demonstrated after repeated assessment participants must be screen failed
* Demonstrated acceptable inhaler use technique for Diskus/Accuhaler (prior to run-in) and Breezhaler (prior to randomization) and able to complete spirometry procedures prior to randomization.
* A parent/legal guardian must be designated to complete all e-Diary entries and attend all clinic visits with the participant.
* Parents/legal guardian must be willing and able to assist the child with the procedures outlined in the protocol, e.g. compliance with study medication, completion of electronic participant diary
* Female participants of child-bearing potential, who might become sexually active, must be informed of the need to prevent pregnancy during the study using effective contraceptive methods. The decision on the contraceptive method should be reviewed at least every 3 months to evaluate the individual need and compatibility of the method chosen.

Exclusion Criteria:

* Systemic corticosteroid use for any reason within 3 months of Run-in
* Participants on low to medium mono ICS alone
* Participants requiring six or more puffs of rescue medication per day on more than two consecutive days in the four weeks prior to Screening (Visit 1) and/or in the four weeks prior to the Run-in visit
* Participants who have had an asthma attack/exacerbation requiring a) systemic corticosteroids (SCS) or b) hospitalization or c) emergency room visit, within 3 months prior to Screening (Visit 1), or more than 3 separate exacerbations in the 12 months preceding the Screening visit
* Participants with a known narrow-angle glaucoma, bladder dysfunction, bladder outlet obstruction or any other conditions where anticholinergic treatment is contraindicated prior to Screening (Visit 1)
* Participants with a history of long QT syndrome or whose corrected QT interval (QTc) measured at start of Run-in and confirmed at Baseline (prior to randomization) (Fridericia method) is prolonged (> 450 msec for boys and girls) and confirmed by a central assessor (these patients should not be rescreened)
* Suspected or documented active infections (bacterial, viral, fungal, mycobacterial or other, including active SARS-CoV-2, tuberculosis or atypical mycobacterial disease) of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 6 weeks of Screening (Visit 1)
* History of Type I diabetes or uncontrolled Type II diabetes
* Participants who are sexually active at screening
* Hemoglobin levels outside normal ranges at Run-in (Visit 20)
* Female patients of childbearing potential (e.g., are menstruating) who do not agree to abstinence or, if they become sexually active during study participation, do not agree to the use of contraception as defined in the inclusion criteria.

Additional protocol-defined inclusion / exclusion criteria may apply.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in trough FEV1 | At the start and end of each 2 week treatment period (Days 1, 14, 29, 42, 57 and 70)
  Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured by spirometry.

SECONDARY OUTCOMES:
Steady state pharmacokinetic (PK) parameters C0 | At the start and end of each 2 week treatment period (Days 1, 14, 15, 29, 42, 43, 57, 70 and 71)
  Steady state pharmacokinetic (PK) parameters C0 will be provided for plasma glycopyrronium concentrations at pre-dose and post-dose time-points.
Systemic exposure following sparse PK sampling | At the start and end of each 2 week treatment period (Days 1, 14, 15, 29, 42, 43, 57, 70 and 71)
  Systemic exposure following sparse PK sampling will be provided at pre-dose and post-dose time-points for each glycopyrronium dose level
Change from Baseline in PEF rate | At the start and end of each 2 week treatment period (Days 1, 14, 15, 29, 42, 43, 57, 70 and 71)
  Morning and Evening Peak Expiratory Flow Rate (PEF) will be measured. PEF is the peak expiratory flow, the maximum speed of expiration.
Change from Baseline in FEV1 | At the start and end of each 2 week treatment period (Days 1, 14, 15, 29, 42, 43, 57, 70 and 71)
  Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured by spirometry.
Change from baseline in rescue medication use | At the start and end of each 2 week treatment period (Days 1, 14, 15, 29, 42, 43, 57, 70 and 71)
  Daily use of rescue medication will be recorded each morning and evening throughout the 2 week treatment by the participant using their electronic diary.
Adverse events of special interest (AESI) typical of anti-muscarinic side effects | From the start of run-in to 30 days after end of treatment, assessed up to maximum duration of 16 weeks
  AESIs that are typical of anti-muscarinic agents will be reported.

CONTACTS AND LOCATIONS:
Locations (22):
- Bulgaria (3):
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sevlievo
  - Novartis Investigative Site, Sofia
- Novartis Investigative Site, Ibagué, Tolima Department, Colombia
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City, GTM
  - Novartis Investigative Site, Guatemala City
- Hungary (6):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Nagykanizsa
  - Novartis Investigative Site, Szigetvár
- Poland (2):
  - Novartis Investigative Site, Tarnów
  - Novartis Investigative Site, Lodz, Łódź Voivodeship
- South Africa (2):
  - Novartis Investigative Site, George, Western Cape
  - Novartis Investigative Site, Cape Town
- Spain (4):
  - Novartis Investigative Site, Esplugues, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Mérida, Extremadura
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.